CLINICAL TRIAL: NCT05848583
Title: A Single-Center, Open-Label Study on the Nutritional Adequacy, Tolerability, and Safety of a Standard Tube Feeding Formula in Adult Participants
Brief Title: Nutritional Tolerance and Safety of a Tube Feeding Formula
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Bruyère Health Research Institute. (Other); Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: N02-20-02-T0005; 23.01.CA.HCN (Other: Sponsor)
Record Dates: First submitted 2023-04-05; First posted 2023-05-08 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Enteral Feeding
Keywords: enteral nutrition; nutrition; gastrointestinal; tube feeding

STUDY DESIGN:
Intervention Model Description: Single center, open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Enteral Nutrition (EN) Formula (Experimental): Enteral formula
  Interventions: Other: Compleat 1.5

INTERVENTIONS:
Other: Compleat 1.5 — EN Formula

SUMMARY:
This open-label, prospective study will be conducted to assess the nutritional efficacy, safety, and tolerance of a concentrated, enteral formula in medically stable adults, who currently require or will require to be enterally fed.

DETAILED DESCRIPTION:
In patients unable to meet energy and protein requirements orally, enteral nutrition (EN) often serves as the sole source of nutrition for long-term tube fed individuals in varied care settings. EN formulas are designed to meet patients' macronutrient needs as well as vitamin and mineral needs with the overall objective of establishing and maintaining quality of life and further preventing undesirable outcomes that are associated with malnutrition. Some individuals who might benefit from a formulation with real food ingredients have not been able to do so because they need a more concentrated, higher calorie formula. Compleat® 1.5 is a calorically dense real food containing nutrition formula. This open-label, prospective study will be conducted to assess the nutritional efficacy, safety, and tolerance of a concentrated, plant-based enteral formula with real food ingredients, Compleat® 1.5, in medically stable adults, who currently require or will require to be enterally fed.

ELIGIBILITY:
Inclusion Criteria:

1. Medically stable, enterally tube-fed adults with a feeding tube diameter of at least 8 French OR medically stable, adults assessed to require enteral feeding initiation with a feeding tube diameter of at least 8 French (2.6 mm).
2. Aged 18 years or older at the time of screening visit.
3. Currently tolerating or determined to tolerate enteral feeding and eligible for feeding with a 1.5 kcal/mL formula, as per PI discretion.
4. Requires or will require enteral tube feeding to provide 90% or more of their daily nutritional needs without the use of modular(s) for at least 14 days.
5. Participant or their Legally Authorized Representatives (LAR) is willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary informed consent (or assent, if capable), carry out all study-related procedures, and communicate effectively with the study staff.

Exclusion Criteria:

1. Has a condition which contraindicates enteral feeding (e.g., intestinal obstruction).
2. Currently using the study formula
3. Any medical condition or contraindicated medications deemed exclusionary by the PI as determined by medical/medication history at the time of screening visit.
4. Any condition, in the opinion of the PI, that would contraindicate use of the study formula (e.g., need for severe fluid restriction, allergy to formula ingredients, etc.).
5. Participation in another interventional clinical study between 30 days prior to screening visit until the end of study.
6. Any condition or abnormality that, in the opinion of the QI, would compromise the safety of the participant or the quality of the study data.
7. Unable to obtain informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Nutritional adequacy (caloric goals) | 14 days
  Daily percentage of caloric nutritional goal met for each participant

SECONDARY OUTCOMES:
Nutritional adequacy (protein intake) | 14 days
  Daily percentage of protein goal met for each participant
Frequency of vomiting | 14 days
  Daily report of frequency of vomiting for each participant
Frequency of abdominal pain | 14 days
  Daily report of frequency of abdominal pain for each participant
Frequency of abdominal distention | 14 days
  Daily report of frequency of abdominal distention for each participant
Frequency of reflux | 14 days
  Daily report of frequency of reflux for each participant
Adverse events Adverse events | 14 days
  Frequency and nature of adverse events (AEs).
Frequency of nausea | 14 days
  Daily report of nausea for each participant
Daily stool description and frequency - Bristol stool scale | 14 days
  Daily stool description and frequency (Bristol stool scale) for each participant

CONTACTS AND LOCATIONS:
Overall Officials: Jean Chouinard, MD, Principal Investigator — Bruyère Health Research Institute.
Locations (1):
- Bruyere Research Institute - Bruyère Continuing Care Complex Care Program - St Vincent Hospital, 60 Cambridge St N, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No